CLINICAL TRIAL: NCT05934734
Title: The Influence of Thoracic Outlet Syndrome Severity on Upper Extremity Function and Neural Integrity: A Cross-Sectional Study
Brief Title: Influence of Thoracic Outlet Syndrome Severity on Upper Extremity Function and Neural Integrity
Status: Completed | Type: Observational
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: 09876543
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Thoracic Outlet Syndrome
MeSH Terms: conditions — Thoracic Outlet Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1 (Mild): Participants with mild self-reported thoracic outlet syndrome symptoms (visual analog scale score 1-3).
  Interventions: Other: No intervention
- Cohort 2 (Moderate): Participants with moderate self-reported thoracic outlet syndrome symptoms (visual analog scale score 4-6). No intervention will be provided.
  Interventions: Other: No intervention
- Cohort 3 (Severe): participants with severe self-reported thoracic outlet syndrome symptoms (visual analog scale score 7-9). No intervention will be provided
  Interventions: Other: No intervention
- Cohort 4 (Very Severe): Participants with very severe self-reported thoracic outlet syndrome symptoms (visual analog scale score 10). No intervention will be provided.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational cross-sectional study. No intervention will be provided. Participants will be assessed and stratified into four cohorts based on self-reported symptom severity of thoracic outlet syndrome using a visual analog scale (VAS) to investigate the relationship between symptom severity and upper extremity function/neural integrity.

SUMMARY:
The purpose of this study is to investigate the relationship between the severity of thoracic outlet syndrome and upper extremity function, as well as neural integrity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Diagnosed with thoracic outlet syndrome
* Willing and able to provide informed consent

Exclusion Criteria:

* History of upper extremity surgery unrelated to thoracic outlet syndrome
* Other upper extremity disorders unrelated to thoracic outlet syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 100 individuals (n=25 per cohort), aged 18-65 years, diagnosed with thoracic outlet syndrome will be recruited for this study. Participants will be recruited from local physical therapy clinics and physician offices. Participants will be screened for eligibility prior to being enrolled in the study and stratified into one of four cohorts based on the severity of self-reported symptoms using a visual analog scale: mild (scores 1-3), moderate (scores 4-6), severe (scores 7-9) and very severe (score 10). Exclusion criteria include a history of upper extremity surgery or other upper extremity disorders not related to thoracic outlet syndrome. All participants will provide written informed consent prior to participating in the study assessments.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Range of Motion (ROM) of the Shoulder joint | Baseline
  Active and passive ROM will be measured using a standard goniometer.
Range of Motion (ROM) of the Elbow joint | Baseline
  Active and passive ROM will be measured using a standard goniometer.
Range of Motion (ROM) of the Wrist joint | Baseline
  Active and passive ROM will be measured using a standard goniometer.
Isometric Muscle Strength of shoulder | Baseline
  Maximum voluntary isometric strength of shoulder muscles will be measured using a handheld dynamometer.
Isometric Muscle Strength of elbow | Baseline
  Maximum voluntary isometric strength of elbow muscles will be measured using a handheld dynamometer.
Isometric Muscle Strength of wrist | Baseline
  Maximum voluntary isometric strength of wrist muscles will be measured using a handheld dynamometer.
Self-reported upper extremity function | Baseline
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire, developed by the Institute for Work and Health, is used to measure patient-reported functional outcomes. The DASH questionnaire consists of 30 questions regarding limitations to complete physical activities due to upper extremity pain/impairment. Participants will be asked to respond to each question based on their experiences over the preceding week according to a 5-point Likert scale ranging from 1 (no difficulty) to 5 (unable to do). Responses will be scored out of 5 and averaged to produce a score out of 100 with higher scores representing greater disability.
Nerve Conduction Studies of ulnar nerve | Baseline
  Nerve conduction studies will assess the function/integrity of the ulnar nerve.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Director — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No